CLINICAL TRIAL: NCT05963529
Title: Evaluating the Validity of a Rapid Humidity Ramp Protocol for Identifying the Upper Environmental Limits of Thermal Compensation in Humans
Brief Title: Validity of Humidity Ramp Protocols for Identifying Limits of Survivability in Heat-exposed Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: uORamp
Record Dates: First submitted 2023-07-13; First posted 2023-07-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Heat Stress; Heat Exposure; Temperature Change, Body; Temperature; Extreme, Exposure
Keywords: Heat wave; Hot weather; Heat strain; Cardiovascular strain; Environmental limits for compensability; Extreme heat events; Heat survivability
MeSH Terms: conditions — Heat Stress Disorders; Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: Each participant will complete four trial conditions including one humidity-ramp protocol and three fixed-condition exposures. The humidity ramp protocol will always be completed first. Ambient temperature will remain constant at 42°C. After a 1-hour equilibrium period, relative humidity will be increased by 3% in 10-min increments, from 28% to 70%. The inflection point for core (esophageal) temperature will be subsequently determined.
  On three separate days following the humidity ramp protocol, participants will complete three fixed-condition exposures in random order: 1) 42°C with relative humidity >5% below the estimate compensability limit (below-threshold condition); 2) 42°C with relative humidity >5% above the estimated compensability limit (above-threshold condition) and 3) 28°C with 35% relative humidity (control condition). Exposure will be terminated early if core temperature exceeds 39.2°C or if the participant requests to withdraw.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be informed of the study interventions before providing informed consent but will be masked to the order the fixed-condition exposures (i.e., participants will not know whether the humidity is above or below their identified inflection point). Data processing and statistical analysis for the fixed-condition exposures will be performed with the analyst blinded to participant and trial conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Humidity-ramp protocol (Other): Healthy male and female volunteers. Participants will complete all exposures. The humidity-ramp protocol will necessarily be performed first. The order of the fixed-condition exposures will be randomized.
  Interventions: Other: Humidity-ramp protocol
- Above-inflection fixed-condition exposure (Experimental): Healthy male and female volunteers. Participants will complete all exposures. The humidity-ramp protocol will necessarily be performed first. The order of the fixed-condition exposures will be randomized.
  Interventions: Other: Above-inflection fixed-condition exposure
- Below-inflection fixed-condition exposure (Experimental): Healthy male and female volunteers. Participants will complete all exposures. The humidity-ramp protocol will necessarily be performed first. The order of the fixed-condition exposures will be randomized.
  Interventions: Other: Below-inflection fixed-condition exposure
- Control fixed-condition exposure (Active Comparator): Healthy male and female volunteers. Participants will complete all exposures. The humidity-ramp protocol will necessarily be performed first. The order of the fixed-condition exposures will be randomized.
  Interventions: Other: Control fixed-condition exposure

INTERVENTIONS:
Other: Humidity-ramp protocol — Participants are exposed to 42°C and 28% relative humidity for 70 minutes. Thereafter, humidity is increased 3% until an ambient humidity of 70% is achieved. The humidity at which esophageal temperature (and rectal temperature and heart rate) inflect is subsequently determined.
  Arms: Humidity-ramp protocol
Other: Above-inflection fixed-condition exposure — After a 1 hour equilibrium at 42°C and 28% relative humidity, humidity will be increased 3% every 10 min until it is ~5% higher than the participants' individual esophageal temperature inflection point identified in the humidity ramp protocol. These conditions will be held constant for the remainder of the 9-hour exposure period (starting from the beginning of equilibrium). Tap water will be provided at regular intervals to limit dehydration.
  Arms: Above-inflection fixed-condition exposure
Other: Below-inflection fixed-condition exposure — After a 1 hour equilibrium at 42°C and 28% relative humidity, humidity will be increased 3% every 10 min until it is ~5% lower than the participants' individual esophageal temperature inflection point identified in the humidity ramp protocol. These conditions will be held constant for the remainder of the 9-hour exposure period (starting from the beginning of equilibrium). Tap water will be provided at regular intervals to limit dehydration.
  Arms: Below-inflection fixed-condition exposure
Other: Control fixed-condition exposure — Participants are exposed for 9-hours to 28°C with 35% relative humidity. Participant will be allowed to drink tap water ad libitum.
  Arms: Control fixed-condition exposure

SUMMARY:
The global populace is at growing risk of heat-related illness due to climate change and accompanying increases in the intensity and regularity of extremely hot temperatures. In heat-exposed persons, heat gain from the environment and metabolism initially exceeds the rate of heat dissipation from the skin. Heat is stored in the body, causing core and skin temperatures to rise, which in turn triggers autonomically mediated elevations in cutaneous blood flow and sweating to facilitate heat loss. If conditions are compensable, heat loss increases until it balances total heat gain. At this point, the rate of heat storage falls to zero (i.e., heat balance is achieved) and body temperature stabilizes, albeit at a level elevated from thermoneutral conditions. If, however, the maximal achievable rate of heat dissipation is insufficient to offset heat gain, conditions are uncompensable, and prolonged exposure will cause a continual rise in core temperature that can compromise health if left unchecked. The environmental limits of compensability (i.e., the temperatures/humidities above which heat balance can not be maintained) are therefore an important determinant of survival during prolonged heat exposure. Evaluating this limit and how it can be modified (e.g., by behavior or individual factors like age or sex) is an increasingly important and active field of study.

Contemporary evaluations of the environmental limits of compensability utilize "ramping protocols" in which participants are exposed to increasing levels of temperature or humidity (in 5-10 min stages) while core temperature is monitored. It is generally observed that core temperature is relatively stable (or rises slightly) in the early stages of exposure but undergoes an abrupt and rapid increase as heat stress becomes more severe. The conditions (e.g., wet-bulb temperature or wet-bulb globe temperature) at this "inflection point" are taken as the limits of compensability. That is, it is assumed that inflection corresponds to the demarcation point, below which core temperature would remain stable for prolonged periods (theoretically indefinitely if hydration is maintained) but above which heat loss is insufficient to offset heat gain, causing core temperature to rise continuously. Despite the increasing use of these protocols, no study has clearly demonstrated their validity for identifying the environmental limits of compensability. The goal of this project is therefore to assess the validity of ramping protocols for determining the ambient conditions above which thermal compensation is not possible.

Enrolled participants will complete four experimental trials in a climate-controlled chamber: one ramping protocol followed by three randomized fixed-condition exposures. In the ramping protocol, participants will rest in 42°C with 28% relative humidity (RH) for 70 min, after which RH will be increased 3% every 10 min until 70% RH is achieved. The core (esophageal) temperature inflection point will be determined. For the fixed-condition exposures, participants will rest in i) 42°C with RH ~5% below their individual inflection point (below-inflection condition), ii) 42°C with RH ~5% above their individual inflection point (above-inflection condition), and iii) 26°C with 45% RH (control condition). Comparing the rate of change in esophageal temperature between each fixed-condition exposure will provide important insight into the validity of ramping protocols for identifying the limits of compensability.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults.
* Aged 18-85 years.
* Non-smoking.
* English or French speaking.
* Ability to provide informed consent.

Exclusion Criteria:

* Physical restriction (e.g., due to disease: intermittent claudication, renal impairment, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis, etc.).
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable (e.g., medications increasing risk of heat-related illness; beta blockers, anticholinergics, etc.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
Esophageal temperature rate of change | End of fixed-condition heat exposure (hour 9 or termination)
  Rate of change of esophageal temperature measured over the final 2-hours of heat exposure
Predicted time until 40.2°C esophageal temperature | End of fixed-condition heat exposure (hour 9 or termination)
  Estimated time for esophageal temperature to reach 40.2°C, a commonly-cited criteria for severe heat-illness (e.g., heat stroke), calculated from the end-exposure esophageal temperature and its rate of change (assuming this rate of change is sustained)
Rectal temperature rate of change | End of fixed-condition heat exposure (hour 9 or termination)
  Rate of change of rectal temperature measured over the final 2-hours of heat exposure
Predicted time until 40.2°C rectal temperature | End of fixed-condition heat exposure (hour 9 or termination)
  Estimated time for rectal temperature to reach 40.2°C, a commonly-cited criteria for

SECONDARY OUTCOMES:
Number of participants unable to finish fixed-condition heat exposure | End of fixed-condition heat exposure (hour 9 or termination)
  Number of participants who could not complete each fixed-condition heat exposure due to participant withdrawal or achieving a core temperature of 39.5°C
Mean skin temperature rate of change | End of fixed-condition heat exposure (hour 9 or termination)
  Rate of change of skin temperature measured over the final 2-hours of heat exposure
Heart rate rate of change | End of fixed-condition heat exposure (hour 9 or termination)
  Rate of change of heart rate measured over the final 2-hours of heat exposure
Esophageal temperature | End of fixed-condition heat exposure (hour 9 or termination)
  Esophageal temperature at the end of the fixed-condition exposures
Rectal temperature | End of fixed-condition heat exposure (hour 9 or termination)
  Rectal temperature at the end of the fixed-condition exposures
Mean skin temperature | End of fixed-condition heat exposure (hour 9 or termination)
  Mean skin temperature at the end of the fixed-condition exposures
Heart rate | End of fixed-condition heat exposure (hour 9 or termination)
  Heart rate at the end of the fixed-condition exposures
Thermal sensation | End of fixed-condition heat exposure (hour 9 or termination)
  Self-reported thermal sensation at the end of the fixed-condition exposures using and 8-point scale ranging from neutral (0) to extremely hot (8).
Sweat rate | End of fixed-condition heat exposure (hour 9 or termination)
  Sweat rate at the end of the fixed-condition exposures (calculated via change in body weight)
Net fluid loss | End of fixed-condition heat exposure (hour 9 or termination)
  Net fluid loss estimated as the percentage change in body mass over the fixed-condition exposures.

OTHER OUTCOMES:
Esophageal temperature inflection point | During the ramp protocol (up to 2.5 hours)
  Inflection point for esophageal temperature during the humidity-ramp protocol
Rectal temperature inflection point | During the ramp protocol (up to 2.5 hours)
  Inflection point for rectal temperature during the humidity-ramp protocol
Heart rate inflection point | During the ramp protocol (up to 2.5 hours)
  Inflection point for heart rate during the humidity-ramp protocol

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Meade, PhD, MPH, Study Director — University of Ottawa; Glen P Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available upon reasonable request and signed access agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available following publication of the primary study report.
Access Criteria: Reasonable request and signed access agreement